CLINICAL TRIAL: NCT00843934
Title: Randomized Controlled Trial of Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma
Brief Title: Trial of Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma
Acronym: ACE500
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Masashi Fujii, Professor, Nihon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE500
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; Trans arterial chemoembolization; Epirubicin; Cisplatin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Epirubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-cancer agent (Experimental)
  Interventions: Drug: epirubicin; Drug: Cisplatin

INTERVENTIONS:
Drug: epirubicin — Arm E: Suspension is prepared before arterial infusion as follows: Epirubicin is dissolved with water-soluble, non-ionized contrast medium then mixed with Lipiodol by pumping. Then this suspension is administered by catheter as quick as possible, and gelatin is infused for arterial embolization. Maximum dose of EPI and Lipiodol are 60mg/m2 and 0.3mL/Kg, respectively.
  Other Names: epi-adriamycin
Drug: Cisplatin — Arm C: Suspension is prepared before arterial infusion as follows: Cisplatin (Water soluble CDDP: IA CALL) is mixed with Lipiodol. Then this suspension is administered by catheter as quick as possible, and gelatin is infused for arterial embolization. Maximum dose of Cisplatin and Lipiodol are 65mg/m2 and 0.3mL/Kg, respectively.
  Other Names: CDDP

SUMMARY:
The purpose of this study is to compare the efficacy and safety of cisplatin (CDDP) and epirubicin (EPI) in the treatment of transcatheter chemoembolization for Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be histologically or clinically proven HCC, inoperable, no indication of local treatment and has measurable lesions.
* Subject must to be the first experience of TACE.
* Subject has no extra-hepatic tumor and no obstruction of main portal vein.
* Subjects must have fully recovered from previous treatment (at least 4 weeks interval is needed from prior chmotherapy or radiation therapy).
* ECOG performance status 0-2
* Child-pugh Class A or B
* Subject must have adequate functions of bonemarrow, renal, circulatory organs and appropriate examination results as below:

  1. Serum Total Bilirubin 2.0mg/mL
  2. WBC 3000/mm3
  3. PLT 50000/mm3
  4. Hb 9.0g/dL
  5. Creatinine ; upper normal limit (UNL)
  6. BUN 25mg/dL
* Written informed consent

Exclusion Criteria:

* Subject has extra hepatic metastasis.
* Tumor thrombosis exists at main portal vein.
* Remarkable artery-portal vein shunt or veno-arterial shunt.
* Uncontrollable ascites or pleural effusion.
* History of severe hypersensitivity.
* Any previous TACE or TAE for HCC.
* Any previous chemotherapy using epirubicin or CDDP.
* Complications as below (except chronic hepatitis or liver cirrhosis)

  1. Severe heart disease
  2. Myocardial infarction within 6 months
  3. Renal insufficiency
  4. Active infections (except virous hepatitis)
  5. Gastrointestinal bleeding
  6. Active double cancer
  7. Hepatic encephalopathy or heavy mental disorder.
* Pregnancy or lactation women, or women with suspected pregnancy or men with willing to get pregnant.
* Any subject judged by the investigator to be unfit for any reason to participate in the study.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
response rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tadatoshi Takayama, M.D., Principal Investigator — Digestive Surgery Nihon University School of Medicine
Locations (1):
- Department of Digestive Surgery, Nihon University School of Medicine, tabashi City, Tokyo, Japan